CLINICAL TRIAL: NCT00399750
Title: A Randomized Prospective Study Comparing Three Regimens of Oxaliplatin Plus Fluoropyrimidine and Avastin for Evaluation of Safety and Tolerability in First-line Treatment of Patients With Advanced Colorectal Cancer.
Brief Title: TREE-2: Three Regimens of Eloxatin in Advanced Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: L_8851
Record Dates: First submitted 2006-11-13; First posted 2006-11-15 (Estimated); Last update posted 2009-10-15 (Estimated); Status verified 2009-10

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Oxaliplatin; Bevacizumab

INTERVENTIONS:
Drug: oxaliplatin
Drug: fluoropyrimidine
Drug: bevacizumab

SUMMARY:
A randomized, controlled, open-label multicenter trial to assess the safety and efficacy of 3 oxaliplatin-fluoropyrimidine containing regimens (mFOLFOX6; bFOL; XELOX) + Bevacizumab (TREE1 and TREE2) as first line therapy of advanced metastatic colorectal cancer.

ELIGIBILITY:
The following information on clinical trials is provided for information purposes only to allow patients and physicians to have an initial discussion about the trial. This information is not intended to be complete information about the trial, to contain all considerations that may be relevant to potential participation in the trial, or to replace the advice of a personal physician or health professional.

INCLUSION CRITERIA:

Subjects must meet all of the following inclusion criteria to be eligible for enrollment into the study:

1. Histologically documented adenocarcinoma of the colon, rectum or appendix.
2. Metastatic/recurrent disease not amenable to potentially curative treatment (e.g., inoperable metastatic disease).
3. No prior chemotherapy for metastatic/recurrent disease. Prior adjuvant treatment with 5-FU/LV and/or IFL is allowed if it is completed at least 6 months before study registration.
4. ECOG Performance Status 0- 1.
5. At least one unidimensionally measurable lesion with a diameter >/= 20 mm using conventional CT or MRI scans or >/= 10 mm using spiral CT scans. If a single lesion is identified as the target lesion, a histological or cytological confirmation of adenocarcinoma is required.
6. Recovery in full from any previous surgical procedure.
7. No other serious concomitant disease.
8. Required baseline laboratory parameters:

   1. Absolute neutrophil count (ANC) >/=1,500/mm3 (standard international [SI] units 109/L);
   2. Platelets >/= 100,000/mm3 (SI units 109/L);
   3. Hemoglobin >/= 8.0 g/dL (SI units mmol/L);
   4. Creatinine </= 1.5 x ULN; Total bilirubin </= 2.0 x ULN;
   5. Serum glutamate-oxalate transferase (SGOT, AST) Serum glutamic pyruvic transaminase (SGPT, ALT) </= 3 x ULN </= 3 x ULN;
   6. Urinalysis - dipstick Protein < +1;
   7. Coagulation PT/PTT (INR) Within Normal Limits for Institution;
   8. Serum pregnancy test for females of childbearing potential: Negative within 7 calendar days of randomization to study

EXCLUSION CRITERIA:

The presence of any of the following will exclude a subject from study enrollment:

1. Prior treatment with oxaliplatin or bevacizumab.
2. Any uncontrolled infection.
3. History of myocardial infarction within the previous 6 months or current clinical evidence of congestive heart failure, non-stable coronary artery disease, clinically significant hypertension (blood pressure of >160/110 mmHg on medication), or symptomatic peripheral vascular disease.
4. History of any other cancer (except non melanoma skin cancer or carcinoma in-situ of the cervix) unless in complete remission and off all therapy for that cancer for at least 5 years.
5. Central nervous system metastases.
6. Peripheral neuropathy of any cause.
7. Pregnant or lactating women.
8. Hypersensitivity to one of the study drugs or ingredients.
9. Participation in any investigational drug study within 4 weeks preceding enrollment.
10. Lack of physical integrity of the upper gastrointestinal tract or malabsorption syndrome.
11. Medical or psychiatric disorders that would interfere with informed consent, compliance or make them a poor risk for participation in this trial.
12. Patients with known DPD deficiency.
13. Patients with interstitial pneumonia or extensive symptomatic fibrosis of the lungs.
14. Patients with calculated creatinine clearance of <30 ml/min using Cockroft and Gault formula.
15. Patients who have received an organ allograft.
16. Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to study entry.
17. Chronic, daily treatment with aspirin (>325 mg/day) or nonsteroidal anti-inflammatory medications (intermittent or "p.r.n." use for pain is permitted).
18. Evidence of a bleeding diathesis or coagulopathy.
19. Subjects found to have proteinuria at baseline - If patients are found to have >/= 1+ proteinuria at baseline screening they should undergo a 24-hour urine collection, which must be an adequate collection and must demonstrate <2g of protein/24 hr to allow participation in the study.
20. Patients on chronic therapeutic Warfarin therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 373
Dates: Start 2002-11; Study Completion 2005-06

PRIMARY OUTCOMES:
To evaluate the safety and efficacy of three oxaliplatin-fluoropyrimidine regimens when combined with bevacizumab as therapy for previously untreated metastatic colorectal cancer (TREE 2)

SECONDARY OUTCOMES:
The overall incidence of grade 3 and grade 4 adverse events during the first 12 weeks of treatment for each of the oxaliplatin-fluoropyrimidine regimens used without bevacizumab (TREE1)
Type, frequency, severity, timing, and relatedness of all adverse events during treatment and for 30 days following discontinuation of treatment for each of the oxaliplatin-fluoropyrimidine regimens when used with or without bevacizumab(TREE1 and TREE2)
Actual treatment administration as characterized by median, mean, and range of doses given; dose modifications, omissions, and delays; and actual and relative dose intensity (TREE1 and TREE2)
Tumor response rate (overall and confirmed) based on application of the Response Evaluation Criteria in Solid Tumors (RECIST) (TREE1 and TREE2)
Time to treatment failure (TTF) (TREE1 and TREE2)
Time to tumor progression (TTP) (TREE1 and TREE2)
Median survival (TREE1 and TREE2)
STUDY DESIGN
A randomized, controlled, open-label multicenter trial to assess the safety & efficacy of 3 oxaliplatin-fluoropyrimidine containing regimens (mFOLFOX6; bFOL; XELOX) +Avastin (TREE1 & TREE2) as first line therapy of advanced metastatic colorectal cancer
Patients enrolled prior to the initiation of Amendment 3 (TREE1) will not be eligible to receive Avastin as a component of their treatment regimen.

CONTACTS AND LOCATIONS:
Overall Officials: Yasir Nagarwala, M.D., Study Director — Sanofi
Locations (1):
- Sanofi-Aventis, Bridgewater, New Jersey, United States